CLINICAL TRIAL: NCT06128681
Title: Application Value of Respiratory Mediastinal Intervention Technique in Diagnosis and Comprehensive Treatment of Diseases
Brief Title: Diagnosis and Comprehensive Treatment of Mediastinal Interventional Technique
Status: Recruiting | Type: Observational
Sponsor: Dan Liu (Other)
Responsible Party: Sponsor-Investigator, Dan Liu, Doctor of Medicine, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Other Study IDs: Tianjinzyyhxkld
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Mediastinal Diseases
MeSH Terms: conditions — Mediastinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mediastinal open group: Mediastinal opening technique was performed with intraairway ultrasound guidance before transbronchial needle biopsy (TBNB). In addition, all patients with active pulmonary sarcoidosis and patients with fibrosing mediastinitis in this group will undergo transbronchial lung biopsy (TBLB) as a standardized supplementary procedure. TBNB and TBLB samples underwent histopathological assessment, single-cell sequencing and other detection methods.
  Interventions: Procedure: Intraairway ultrasound-guided mediastinal opening technique; Procedure: Transbronchial Lung Biopsy (TBLB)
- Non-mediastinal open group: Diagnosis are routinely performed without mediastinal opening technique before transbronchial needle biopsy (TBNB).In addition, all patients with active pulmonary sarcoidosis and patients with fibrosing mediastinitis in this group will undergo transbronchial lung biopsy (TBLB) as a standardized supplementary procedure.TBNB and TBLB samples underwent histopathological assessment, single-cell sequencing and other detection methods.
  Interventions: Procedure: Transbronchial Lung Biopsy (TBLB)

INTERVENTIONS:
Procedure: Intraairway ultrasound-guided mediastinal opening technique — Mediastinal intervention for patients with mediastinal imaging abnormalities is performed under general anesthesia to obtain biopsy specimens for detection or elimination of mediastinal masses
  Groups: Mediastinal open group
Procedure: Transbronchial Lung Biopsy (TBLB) — A standardized supplementary procedure performed in all patients with active pulmonary sarcoidosis and fibrosing mediastinitis, regardless of their primary study group assignment, to obtain lung tissue for histopathological diagnosis and disease activity assessment.

SUMMARY:
The goal of this observational study is to learn whether patients undergoing mediastinal disease diagnosis and combined treatment with intrapacial ultrasound-guided mediastinal opening techniques have greater clinical benefit.

The main questions it aims to answer are:

* Whether the mediastinal ultrasound-guided mediastinal opening technique is more beneficial for the diagnosis of benign or malignant mediastinal diseases.
* Does the mediastinal ultrasound-guided mediastinal opening technique benefit the patient by ablating mediastinal masses using freezing, laser, or other means.

Mediastinal diseases were diagnosed by lymph node biopsy combined with NGS, ROSE and other techniques using transairway ultrasound-guided mediastinal opening technique. Ablation of mediastinal malignancies is performed using techniques such as freezing or laser. Transbronchial lung biopsy(TBLB) may also be performed when necessary. Researchers will compare the experimental group with mediastinal opening and the control group without mediastinal opening to see if Mediastinal open technique benefits patients.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic abnormalities of mediastinum
* Can tolerate general anesthesia
* Can tolerate bronchoscopy and has the condition to have mediastinal biopsy and treatment

Exclusion Criteria:

* Imaging or other tests can make a definitive diagnosis
* Cannot tolerate general anesthesia or tracheoscopic surgery
* Patients cannot sign informed consent forms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient had mediastinal imaging abnormalities, and the disease type could not be identified through routine examination, and it was difficult to carry out further treatment or the patient was not satisfied with the previous treatment effect; In addition, patients with clearly diagnosed malignant tumors are difficult to perform tumor resection, or patients with other reasons are difficult to tolerate surgical open surgery, and mediastinal tumor ablation can reduce tumor compression and achieve the purpose of tumor reduction
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
In the diagnosis of mediastinal diseases, the difference in diagnosis rate between the experimental group with open mediastinum and the control group with traditional methods was observed | 11 months
  The contribution of pathological results to the final diagnosis of the disease between the experimental group and the control group was observed.That is, the difference in diagnostic accuracy between the experimental group and the control group.

SECONDARY OUTCOMES:
Overall Survival | 11 months
quality of life survey | 11 months
number of hospitalizations | 11 months
Cost of disease treatment | 11 months

OTHER OUTCOMES:
Immune cell profiling via single-cell RNA sequencing | At the time of biopsy and sample collection
  Single-cell RNA sequencing will be performed on blood, bronchoalveolar lavage fluid (BALF), transbronchial needle biopsy (TBNB) and transbronchial lung biopsy (TBLB) tissue samples to characterize immune cell profiles, identify pathogenic mechanisms, and discover potential therapeutic targets in patients with active pulmonary sarcoidosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China